CLINICAL TRIAL: NCT03572296
Title: Effect of Drinks Containing Fruit Polyphenol Extracts and Fibre on Postprandial Glycaemia. The Glu-MIX Study
Brief Title: Effect of Drinks Containing Fruit Polyphenol Extracts and Fibre on Postprandial Glycaemia. (Glu-MIX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucozade Ribena Suntory (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HVS-010
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Postprandial Period
Keywords: Blackcurrant; Polyphenols; Pulp; Fibre; Glucose; Postprandial; Metabolism; Cognition
MeSH Terms: interventions — Polyphenols; Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Cross-over design. Each participant receives placebo plus 2 treatments.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): No polyphenols or fibre will be delivered in a low sugar drink.
  Interventions: Dietary Supplement: Placebo
- Polyphenol and fibre (Experimental): Blackcurrant extract (800 mg total polyphenols) and pulp (source of fibre) will be delivered in a low sugar drink.
  Interventions: Dietary Supplement: Polyphenol and fibre
- Fibre (Experimental): Pulp (source of fibre) will be delivered in a low sugar drink.
  Interventions: Dietary Supplement: Fibre

INTERVENTIONS:
Dietary Supplement: Placebo — Drinks will be delivered in random order at 3 separate study visits immediately before a high carbohydrate meal. A minimum of 4 days (ideally 7 days) wash-out period will be required between study days.
  Arms: Placebo
Dietary Supplement: Polyphenol and fibre — Drinks will be delivered in random order at 3 separate study visits immediately before a high carbohydrate meal. A minimum of 4 days (ideally 7 days) wash-out period will be required between study days.
  Arms: Polyphenol and fibre
Dietary Supplement: Fibre — Drinks will be delivered in random order at 3 separate study visits immediately before a high carbohydrate meal. A minimum of 4 days (ideally 7 days) wash-out period will be required between study days.
  Arms: Fibre

SUMMARY:
Postprandial glycaemia refers to the transient rise in blood glucose levels that occurs after consuming a meal. Large fluctuations in blood glucose levels, experienced on a frequent basis, may impair the functioning of pancreatic beta cells, and thus elevate the risk of developing type 2 diabetes mellitus (T2DM) and cardiovascular disease. Our group has previously shown that consuming a drink containing fruit polyphenols immediately before a meal, may reduce postprandial glycaemia. Importantly, other fruit components, namely soluble fibres, also impact on carbohydrate digestion by slowing gastric emptying rates. Combining fruit polyphenols and fibre in a drink may, potentially, have additive or synergistic effects on reducing postprandial glycaemia.

This study will investigate the effects of drinks containing blackcurrant polyphenol extract combined with pulp (source of fibre), and pulp alone, on postprandial outcomes and cognitive function following a mixed carbohydrate (starch and sucrose) test meal.

DETAILED DESCRIPTION:
Intake of carbohydrate-rich foods transiently increases blood glucose levels (known as postprandial glycaemia). Repeated, high, postprandial glucose responses are evidenced to impair pancreatic beta cell function, thus increasing the risk of developing type-2 diabetes mellitus and cardiovascular disease. Therefore, meals that elicit a reduced, or more gradual, rise in blood glucose levels are desirable.

Previous studies have shown that consuming a drink containing fruit polyphenols, such as those from blackcurrants (BC), immediately before a high carbohydrate meal, reduced the postprandial glycaemic response. Importantly, other fruit components, namely soluble fibres, also impact on carbohydrate digestion by slowing gastric emptying rates. It is not yet known the effect of combining fibre and polyphenols on postprandial glycaemia. Although limited, there is a growing body of evidence showing beneficial acute effects of polyphenols in cognitive function which is of great interest in many work and academic environments where fast cognitive enhancement is wanted to perform a task or an exam.

This study will investigate the effects of drinks containing BC polyphenol extract combined with pulp (source of fibre), and pulp alone, on postprandial outcomes and cognitive function following a mixed carbohydrate (starch and sucrose) test meal.

Study design: A randomised, controlled, double-blind, cross-over study, of the healthy adult UK population, will be conducted. All subjects will receive the placebo drink, pulp only drink and the pulp with polyphenol drink in a random order. Baseline (fasted) blood samples will be taken before consuming the test drink (T0 min). Immediately following consumption of the drink, a mixed carbohydrate test meal will be consumed. Further blood samples will be collected at regular times until T150 min. Blood samples will be analysed for plasma glucose, insulin, glucose-dependent insulinotropic peptide (GIP) and C-peptide. Subjects will also perform a 30 min computer based cognitive performance test at baseline (T-45 min) and endpoint (T165 min). Visual analogue scales will be used to assess the effect of the test drinks on a range of sensory characteristics e.g. palatability, satiety and subjective mood feelings. Finally, an ad libitum pasta meal at the end of the study visit (T 215 min) will be used to assess the effects on energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Men and women
* Healthy (free of diagnosed diseases listed in the exclusion criteria)
* Body Mass Index 18-35 kg/m2
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Those diagnosed with Phenylketonuria (PKU)
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breastfeeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months.
* Full Blood Counts and Liver Function test results outside of the normal range.
* Current smokers, or reported giving up smoking within the last 6 months
* History of substance abuse or alcoholism
* Reported history of Cardiovascular disease, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function
* Unwilling to restrict consumption of specified high polyphenol/ high fibre foods for 48 h before the study
* Weight change >3 kg in preceding 2 months
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.5 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study: alpha-glucosidase inhibitors (acarbose: Glucobay), insulin sensitizing drugs (metformin: Glucophage, Glucophage SR, Eucreas, Janumet; thiazolidinediones: Actos, Competact), sulfonylureas (Daonil, Diamicron, Diamicron MR, Glibenese, Minodiab, Amaryl Tolbutamide), and lipid lowering drugs (statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates). Other medications should be reviewed by medical representative from KCL on a case by case basis.
* Nutritional supplements that may interfere with the study: higher dose vitamins/minerals (>200% Recommend Nutrient Intake), B vitamins, Vitamin C, calcium, copper, chromium, iodine, iron, magnesium, manganese, phosphorus, potassium and zinc. Subjects already taking vitamin or minerals at a dose around 100% or less up to 200% of the RNI, or evening primrose/algal/fish oil supplements will be asked to maintain habitual intake patterns, ensuring that they take them every day and not sporadically. They will be advised not to stop taking supplements or start taking new supplements during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemia (iAUC 0-30 min) | 30 min
  The primary endpoint is iAUC 0-30 min for plasma glucose concentrations

SECONDARY OUTCOMES:
Postprandial glycaemia: iAUC 0-120 min | 120 min
  iAUC 0-120 min for plasma glucose concentrations
Postprandial glycaemia: iAUC 0-150 min | 150 min
  iAUC 0-150 min for plasma glucose concentrations
Postprandial glycaemia: iCmax | 150 min
  iCmax for plasma glucose concentrations
Postprandial glycaemia: Tmax | 150 min
  Tmax for plasma glucose concentrations
Postprandial glycaemia: absolute concentrations at specific time points | 150 min
  Absolute concentrations at specific time points, for plasma glucose concentrations
Postprandial insulinemia: iAUC 0-30 min | 30 min
  iAUC 0-30 min for serum insulin concentrations
Postprandial insulinemia: iAUC 0-120 min | 120 min
  iAUC 0-120 min for serum insulin concentrations
Postprandial insulinemia: iAUC 0-150 min | 150 min
  iAUC 0-150 min for serum insulin concentrations
Postprandial insulinemia: iCmax | 150 min
  iCmax, for serum insulin concentrations
Postprandial insulinemia: Tmax | 150 min
  Tmax for serum insulin concentrations
Postprandial insulinemia: absolute concentrations at specific time points | 150 min
  Absolute concentrations at specific time points, for serum insulin concentrations
Postprandial C-peptide: iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma C-peptide concentrations
Postprandial C-peptide: iAUC 0-120 min | 120 min
  iAUC 0-120 min for plasma C-peptide concentrations
Postprandial C-peptide: iAUC 0-150 min | 150 min
  iAUC 0-150 min for plasma C-peptide concentrations
Postprandial C-peptide: iCmax | 150 min
  iCmax for plasma C-peptide concentrations
Postprandial C-peptide: Tmax | 150 min
  Tmax for plasma C-peptide concentrations
Postprandial C-peptide: Absolute concentrations at specific time points | 150 min
  Absolute concentrations at specific time points, for plasma C-peptide concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iAUC 0-120 min | 120 min
  iAUC 0-120 min for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iAUC 0-150 min | 150 min
  iAUC 0-150 min for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iCmax | 150 min
  iCmax, for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): Tmax | 150 min
  Tmax for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): Absolute concentrations at specific time points | 150 min
  Absolute concentrations at specific time points, for plasma GIP concentrations
Cognitive function test scores | Before and after 150 min blood collection
  Descriptive statistics

OTHER OUTCOMES:
7-d food diary (estimated/unweighed) | 7-days
  Habitual dietary intake analysis
100 mm visual analogue scale (VAS) measures of the palatability of the study drink | 10 min following the test drink
  For each VAS, a numerical score between 0 (not at all) and 100 (extremely) mm was obtained.
100 mm visual analogue scale (VAS) measures of mood, satiety and digestive comfort | 150 min
  For each VAS, a numerical score between 0 (not at all) and 100 (extremely) mm was obtained.
Ad libitum energy intake | 15 min
  Energy intake during ad libitum meal
100 mm visual analogue scale (VAS) measures of the palatability of the ad libitum meal | 15 min following the ad libitum meal
  For each VAS, a numerical score between 0 (not at all) and 100 (extremely) mm was obtained.
Buccal mouth swab | One off sample, collected at the first 1 day of study visit
  Future exploratory analysis of lactase activity via the derived allele at the European

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Metabolic Research Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Acosta ML, Smith L, Miller RJ, McCarthy DI, Farrimond JA, Hall WL. Drinks containing anthocyanin-rich blackcurrant extract decrease postprandial blood glucose, insulin and incretin concentrations. J Nutr Biochem. 2016 Dec;38:154-161. doi: 10.1016/j.jnutbio.2016.09.002. Epub 2016 Sep 14. PMID 27764725
- [Derived] Pinto AM, Hobden MR, Brown KD, Farrimond J, Targett D, Corpe CP, Ellis PR, Todorova Y, Socha K, Bahsoon S, Haworth C, Marcel M, Nie X, Hall WL. Acute effects of drinks containing blackcurrant and citrus (poly)phenols and dietary fibre on postprandial glycaemia, gut hormones, cognitive function and appetite in healthy adults: two randomised controlled trials. Food Funct. 2023 Nov 13;14(22):10163-10176. doi: 10.1039/d3fo03085g. PMID 37902089